CLINICAL TRIAL: NCT07285733
Title: Multimodal Neuromonitoring at the ICU
Acronym: NEMO-RETRO
Status: Completed | Type: Observational
Sponsor: University Hospital, Antwerp (Other)
Collaborators: CENTER TBI (Unknown); Research Foundation - Flanders (Fonds Wetenschappelijk Onderzoek) (Other)
Responsible Party: Principal Investigator, Philppe Jorens, MD, PhD, University Hospital, Antwerp
Other Study IDs: EDGE 4584
Record Dates: First submitted 2025-11-19; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-11

CONDITIONS: Traumatic Brain Injury; Subarachnoid Aneurysm Hemorrhage
Keywords: Neuromonitoring
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Cerebrospinal fluid and plasma were retained in the original prospective study. No additional biospecimens will be included in this retrospective study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute brain injury: Patients with acute brain injury (TBI or aSAH)
  Interventions: Device: Multimodal neuromonitoring

INTERVENTIONS:
Device: Multimodal neuromonitoring — Imaging: CT, MRI, XA Neuromonitoring: Brain Tissue Monitoring Probe, Hemedex, External ventricular drain, Cortical microdialysis catheter Other monitoring: Arterial catheter, Jugular bulb catheter, routine vital parameters

SUMMARY:
Neurocritical care has become a distinct discipline within the field of intensive care medicine with a major focus on the treatment of patients with acute damage to the most complex organ of the human body, the brain. The main indications for acute neurocritical care concern aneurysmal Subarachnoid Hemorrhage (SAH) and severe Traumatic Brain Injury (TBI). These disease entities form a major health and socioeconomic problem as they afflict young patients and the rate of death and disability is high. The pathology and treatment of these patients is heterogeneous and complex. Despite advances in basic neuroscience which have increased our understanding of processes in the injured brain, approaches to management are largely unfocused and adhere to the concept of a 'one pill for everybody' approach. Novel monitoring technology and new neuroimaging techniques now offer opportunities for advancing the care for these patients to a more individualized targeted management.

In the period of 2010-2014, a prospective trial was conducted in the Antwerp University Hospital, including 50 patients with either SAH or TBI, who underwent extensive monitoring, known as "Individualized targeted management in neurocritical care".

In NEMO-RETRO, the investigators want to answer proposed and new research questions in retrospective analyses, using current insights and methodologies.

Objectives:

1. Cerebral blood flow monitoring

   1. Investigate the effect of changes in therapy (nature/intensity) on Cerebral Blood Flow (CBF) measured by thermal diffusion flowmetry and Transcranial Doppler (TCD)
   2. Determine the added value of continuous CBF monitoring for the early detection of vasospasm and ischaemia
2. Brain tissue oxygen tension

   1. Investigate the effect of changes in therapy (nature/intensity) on cerebral oxygenation as measured by Brain Tissue Oxygen Tension (PTiO2)
   2. Investigate the relation between PTiO2 and hemodynamic parameters such as CBF, CPP, and ICP
3. Systemic effects of brain specific therapy

   1. Investigate the effects of brain-targeted therapy on cardiac output and lung function
   2. Determine the relation of CBF to cardiac output, in particular following triple H therapy
4. Neuroimaging

   1. Accurately document structural brain damage following TBI and SAH
   2. Document vasospasm and quantify flow and perfusion
   3. Quantify the degree of secondary ischaemic damage to the brain
   4. Differentiate swelling from edema
   5. Train and validate models to interpret neuroimaging
5. Outcome

   1. Assess global functional outcome at 6 months post-injury
   2. Assess health-related quality of life at 6 months after injury
6. Integrated approach analysis

   1. Describe the effects of brain-targeted therapy on cerebral and systemic parameters
   2. Define the added value of extended multimodality monitoring and advanced neuroimaging to detect vasospasm and secondary ischaemic damage, defined by markers of neuronal injury and cell death
   3. Develop recommendations for individualized targeted management

ELIGIBILITY:
This study is based on the 50 patients recruited for the original study.

For TBI:

Inclusion Criteria:

* male or female patients aged 18 to 70 years, inclusive
* sustained head injury within the previous 24 hours
* TBI diagnosed by history, clinical examination with a GCS of 12 or less
* evidence of TBI confirmed by abnormalities on CT scan
* clinical indication to monitor ICP
* informed consent is obtained from the patient or from a legally acceptable representative

Exclusion Criteria:

* life expectancy of less than 24 hours as determined by the investigator
* any spinal cord injury
* coma suspected to be primarily due to causes other than head injury, such as drug or alcohol overdose
* clinically significant or active gastro-intestinal, renal, hepatic, endocrine or CNS disease or chronic condition (e.g.psychiatric disorder) that can be ascertained at the time of admission and could affect functional outcome
* respiratory/hemodynamic instability, refractory to treatment and precluding transport for neuroimaging studies
* pregnancy
* special exclusion criteria for MRI, such as non-removable metals, artificial joints, electronic devices (pacemaker, pumps etc.)
* informed consent is obtained from a legally acceptable representative, prior to any study related activity

For aneurysmal subarachnoid hemorrhage:

Inclusion Criteria:

* male or female patients aged 18 to 70 years, inclusive
* ruptured aneurysm, demonstrated by CT angiography or DSA
* onset of SAH clinical symptoms within the preceding 72 hours
* World Federation of Neurosurgery (WFNS) grade III-IV and grade V patients, who improve within 24 hours after ventriculostomy
* indication for ICP monitoring or CSF drainage
* informed consent is obtained from the patient or a legally acceptable representative

Exclusion Criteria:

* non-aneurysmal subarachnoid hemorrhage
* admission in a clinical state with extremely poor prognosis (e.g. wide, non-reactive pupils for more than 1 hour)
* significant coagulation disturbances (thrombocytes < 80 per mL, partial thromboplastin time > 45 sec, INR > 1.5)
* cytostatic therapy in patients with malignant disease
* pregnancy
* special exclusion criteria for MRI, such as non-removable metals, artificial joints, electronic devices (pacemaker, pumps etc.)
* respiratory and/or hemodynamic instability precluding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primarily admitted to the Antwerp University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2010-02 (Actual); Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Number of participants with a favourable neurological outcome | From enrollment to the end of follow-up at 6 months
  Glasgow Outcome Scale - Extended (GOSE; 1 = Dead, 8 = Upper good recovery)

SECONDARY OUTCOMES:
Change from baseline in abnormalities on neuroimaging through CT, MRI or XA | From enrollment to the end of the study at 6 months
  Change based on evolution of bleeding areas, ischemic areas, edema

OTHER OUTCOMES:
Change from baseline in NSE | From enrollment up to 12 days, unless earlier ICU discharge
  Measurement of neuron-specific enolase (ng/mL, plasma/CSF)
Change from baseline in GFAP | From enrollment up to 12 days, unless earlier ICU discharge
  Measurement of glial fibrillary acidic protein (ng/mL, plasma/CSF)
Change from baseline in S100B | From enrollment up to 12 days, unless earlier ICU discharge
  Measurement of S100 calcium-binding protein B (ng/mL, plasma/CSF)
Change from baseline in NFL | From enrollment up to 12 days, unless earlier ICU discharge
  Measurement of neurofilament light chain (ng/mL, plasma/CSF)
Change from baseline in UCH-L1 | From enrollment up to 12 days, unless earlier ICU discharge
  Measurement of ubiquitin carboxy-terminal hydrolase L1 (ng/mL, plasma/CSF)
Change from baseline in MDA | From enrollment up to 12 days, unless earlier ICU discharge
  Measurement of malondialdehyde (µmol/L)
Change from baseline in Ferritin | From enrollment up to 12 days, unless earlier ICU discharge
  Measurement of ferritin (ng/mL)
Change from baseline in Hepcidin | From enrollment up to 12 days, unless earlier ICU discharge
  Measurement of hepcidin (ng/mL)
Change from baseline in GDF-15 | From enrollment up to 12 days, unless earlier ICU discharge
  Measurement of growth differentiation factor 15 (ng/mL)
Change from baseline in CHI3L1 | From enrollment up to 12 days, unless earlier ICU discharge
  Measurement of chitinase-3-like protein 1 (ng/mL)
Change from baseline in TfR | From enrollment up to 12 days, unless earlier ICU discharge
  Measurement of transferrin receptor (ng/mL)
Change from baseline in IL-1α | From enrollment up to 12 days, unless earlier ICU discharge
  Measurement of interleukin-1 alpha (pg/mL)
Change from baseline in Fe²⁺ | From enrollment up to 12 days, unless earlier ICU discharge
  Measurement of ferrous iron (µmol/L)
Change from baseline in Syndecan | From enrollment up to 12 days, unless earlier ICU discharge
  Measurement of syndecan (ng/mL)
Change from baseline in IL-1β | From enrollment up to 12 days, unless earlier ICU discharge
  Measurement of interleukin-1 beta (pg/mL)
Change from baseline in IL-6 | From enrollment up to 12 days, unless earlier ICU discharge
  Measurement of interleukin-6 (pg/mL)
Change from baseline in IL-10 | From enrollment up to 12 days, unless earlier ICU discharge
  Measurement of interleukin-10 (pg/mL)
Change from baseline in IL-18 | From enrollment up to 12 days, unless earlier ICU discharge
  Measurement of interleukin-18 (pg/mL)
Change from baseline in IL-23 | From enrollment up to 12 days, unless earlier ICU discharge
  Measurement of interleukin-23 (pg/mL)
Change from baseline in IL-1RA | From enrollment up to 12 days, unless earlier ICU discharge
  Measurement of interleukin-1 receptor antagonist (pg/mL)
Change from baseline in TNFα | From enrollment up to 12 days, unless earlier ICU discharge
  Measurement of tumor necrosis factor alpha (pg/mL)

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be shared in accordance with the defined research questions. All data will be anonymized prior to analysis, and transfer procedures will be carried out in full compliance with hospital regulations.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months and ending 1 year after publication of results.
Access Criteria: Researchers may request data by contacting the original investigators. An official application must be submitted to the original investigators, who will determine whether data sharing is approved. In the event of approval, a formal data-sharing agreement will be established between the requesting researchers and the original investigators. All data sharing will be conducted in accordance with the local regulations of Antwerp University Hospital.